CLINICAL TRIAL: NCT05515575
Title: Phase II Study of Niraparib in Soft Tissue Sarcoma Patients With Altered DNA Damage Repair
Brief Title: A Study of Niraparib in People With Soft Tissue Sarcoma Who Have Changes in Their Tumor DNA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-089
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Sarcoma,Soft Tissue; Sarcoma Uterus
Keywords: Niraparib; 22-089
MeSH Terms: conditions — Sarcoma | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: This will be a single-center, open label, phase II study of niraparib and will utilize Simon's two-stage design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib (Experimental): This study will utilize Simon's two-stage design: 16 patients will be enrolled in the first portion of this study. If 4 or more patients are progression-free at 12 weeks, an additional 16 patients will be enrolled for a total of n = 32 patients enrolled.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Each patient will receive niraparib daily in 21-day cycles until disease progression or unacceptable toxicity. Mandatory baseline tumor biopsies will occur during study screening, if feasible.

SUMMARY:
The purpose of this study is to test whether the study drug, niraparib, is effective against unresectable and/or metastatic soft tissue sarcoma with DDR mutations. The researchers will also study whether niraparib is safe and causes few or mild side effects, and whether there are groups of DDR mutations in soft tissue sarcoma cells that respond better to treatment with niraparib.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent
* Participants or their legally authorized representatives (LARs) need to be willing to provide written informed consent/assent for the trial
* Be willing to comply with treatment protocol
* Histologically confirmed unresectable or metastatic soft tissue or uterine sarcoma
* Known deleterious or suspected deleterious alteration in at least one of the following prespecified DDR pathway genes:

Core Genes

Gene Pathway

BRCA1 FA/HR

BRCA2 FA/HR

BRIP1 FA/HR

BARD1 FA/HR

BLM FA/HR

PALB2 FA

MRE11 HR

NBN HR

RAD50 HR/NHEJ

RAD51B FA/HR

RAD51C HR

RAD51D HR

RAD52 HR

RAD54B HR

Other Genes

Gene Pathway

ABRAXAS1 NHEJ

ATM OTHER

ATR OTHER

CHEK1 OTHER

CHEK2 OTHER

ERCC4 NER

ERCC8 NER

FANCA FA

FANCC FA

FANCD2 FA

FANCE FA

FANCF FA

FANCG FA

FANCI FA

FANCL FA

FANCM FA/HR

MDC1 OTHER

PARP1 BER

RAD23B NER

RECQL4 HR

RPA1 NER

SLX4 FA/HR

XRCC2 FA/HR

XRCC4 NHEJ

XRCC6 NHEJ

A= Fanconi Anemia BER = Base Excision Repair NER = Nucleotide Excision Repair HR = Homologous Recombination NHEJ = Non-homologous End Joining

* Additional genes may be added to Appendix 18.1 in a study addendum as medical and scientific research and/or diagnostic testing evolves
* Alterations of uncertain significance must be approved for inclusion by the Principal Investigator

  * Performance status of ECOG ≤ 2
  * Progressed on at least 1 prior line of systemic therapy.
* Patients who decline standard of care first-line systemic therapy will be permitted to enroll
* Prior adjuvant therapy will not count if it was completed more than 1 year before the date of consent

  * Presence of measurable disease by RECIST 1.1
* Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment.

  * Adequate organ function determined within 14 days of treatment initiation, defined below:
* Absolute neutrophil count (ANC) ≥ 1.5 K/mcL
* Platelets ≥ 100 K/ mcL
* Hemoglobin ≥ 9 g/dL
* Serum creatinine OR Measured or calculated creatinine clearance Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 . For calculated CrCL, the Cockcroft Gault formula or institutional standard formula can be used.
* Serum total bilirubin ≤1.5 X ULN OR ≤2 X ULN if hyperbilirubinemia is due to Gilbert's syndrome
* AST (SGOT) and ALT (SGPT) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN); if liver metastases, then ≤ 5 × ULN
* International Normalized Ratio ≤1.5 X ULN (≤ 2.5 × ULN if on anticoagulants)

  * Women of childbearing potential must have a negative serum pregnancy test at screening and ≤ 72 hours prior to the first dose of study treatment.
  * Women of childbearing potential must be willing to use a highly effective method of contraception and not breastfeed for the duration of the study and for at least 6 months after the last dose of study medication
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

  * Non-sterile male subjects and their female partners must be willing to use a highly effective method of contraception during the study treatment period and for at least 3 months after the last dose of study treatment. Nonsterile males must avoid sperm donation for the duration of the study and for at least 3 months after last study drug.
  * Prior chemotherapy or any investigational therapies or other anti-cancer agent must have been completed at least 4 weeks before the study drug administration. All AEs must be ≤ NCI CTCAE v5 Grade 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline. Patients who were treated with estrogen modulating therapies (aromatase inhibitors, tamoxifen, GnRH agonists etc.) must have been treated at least 2 weeks prior to study drug administration.
  * Radiation therapy encompassing >20% of the bone marrow is prohibited within 2 weeks prior to Day 1 and during study treatment. Note: Palliative radiation therapy to a small field >1 week prior to Day 1 of study treatment may be allowed.
  * Patients must have normal blood pressure or adequately treated and controlled hypertension. (i.e. systolic BP ≤ 140 mmHg and diastolic BP ≤ 90 mmHg) .
  * Patients receiving corticosteroids may continue as long as their dose is stable for at least 4 weeks prior to initiating protocol therapy.
  * Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with documented undetectable viral load and CD 4 count ≥350 within 6 months of the first dose of study treatment are eligible for this trial.

Exclusion Criteria:

* Patient is simultaneously enrolled on any therapeutic clinical trial.
* Patient has had major surgery within 3 weeks prior to initiating protocol therapy. Note: patient must have recovered from any surgical effects.
* Uncontrolled intercurrent illness including current active or chronic infection requiring systemic therapy or the following cardiac criteria:

  * Symptomatic congestive heart failure (NYHA classification III or IV) within 6 months
  * Acute myocardial infarction ≤6 months prior to Day 1
  * Grade ≥2 ventricular arrhythmia ≤6 months prior to Day 1
  * History of cerebrovascular accident within 6 months before first dose of study drugs
* Participant has leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiologic signs of CNS hemorrhage.

Note: Participants with asymptomatic brain metastases (i.e. off corticosteroids and anticonvulsants for at least 7 days) are permitted.

* Known history of active Mycobacterium tuberculosis infection
* Prior therapy with a PARP inhibitor
* Patients who have not recovered from clinically significant adverse events of prior therapy to ≤ NCI CTCAE v5 Grade 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline.

  °If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy events due to a previously administered agent.
* Presence of a gastrointestinal condition that may affect drug absorption
* Known allergy or reaction to any component of the study drug or its excipients.
* Women who are pregnant or breast feeding
* Patients expecting to have a child within the projected duration of the trial, starting with the pre-screening or screening visit through 6 months after the last dose of study treatment(s) for women or 7 months for men.
* Prior allogeneic stem cell transplantation or organ transplantation.
* Participant has received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* Participant has received colony stimulating factors (e.g., granulocyte colonystimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.

  °If growth factors were used as neutropenic fever prophylaxis during a previous treatment regimen then enrollment is allowed, as long as 2 weeks as elapsed from the prior dose
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Participant has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Participant has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).

  * Patients with chronic HBV infection with active disease who are on suppressive antiviral therapy prior to initiation of cancer therapy
  * Patients with HCV on treatment are eligible if HCV viral load is below the level of quantification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 12 weeks
  Defined by RECIST 1.1. PFS is defined as the period from start of study treatment until recurrent or progressive of disease (POD) is objectively documented (taking as reference for progressive disease the smallest measurement recorded on study), death, or date of last study visit involving assessment of disease status.

SECONDARY OUTCOMES:
Assess adverse events | 2 years
  as defined by CTCAE v 5.0
Progression free survival (PFS) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sujana Movva, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm